CLINICAL TRIAL: NCT04996199
Title: Comparative Efficacy of Carbamazepine Versus Oxcarbazepine in Treatment of Trigeminal Neuralgia- a Randomized Controlled Clinical Study
Brief Title: Comparision Efficacy of Carbamazepine & Oxcarbazepine in the Treatment of Trigeminal Neuralgia- a Randomised Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: suman008
Record Dates: First submitted 2020-03-21; First posted 2021-08-09 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-08

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Oxcarbazepine; Carbamazepine; zileuton

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxcarbazepine GROUP (Experimental): Oxcarabazepine 150mg BD starting dose & will be increased if the patient is not relieved
  Interventions: Drug: Oxcarbazepine
- Carbamzepine GROUP (Active Comparator): carbamazepine 100mg BD initial dose & will be increased if the patient is not relieved
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Oxcarbazepine — oxcarbazepine 150mg BD initial dose , followup will be done at 15days, 6weeks, 10 weeks interval
  Other Names: LOVAX
  Arms: Oxcarbazepine GROUP
Drug: Carbamazepine — carbamazepine 100mg BD initial dose, follow up will be done 2weeks, 6 weeks & 10weeks
  Other Names: zileuton
  Arms: Carbamzepine GROUP

SUMMARY:
Trigeminal neuralgia is a neuropathic facial pain condition, characterized by unilateral paroxysmal pain which can be described as stabbing or electric shock like, in the distribution of one or more divisions of trigeminal nerve which is triggered by innocuous stimuli. The attack is provoked by touching or stimulating these trigger zones. There are various pharmacological drugs present for the treatment of trigeminal neuralgia. Carbamazepine and oxcarbazepine are the first-choice drugs for the treatment of TN. Other drugs include lamotrigine , baclofen , gabapentin, antidepressants , eslicarbazepine , sumatriptan & vixitrigine. The carbamazepine is first choice of drug which has serious side effects including dizziness, memory loss, sleppiness, aplastic anaemia. Oxcarbazepine has similar mechanism of action and found to have lesser adverse events when used in various neuralgias in the place of carbamazepine. But there is still lack of evidence to prove that oxcarbazepine can be used as monotherapy in TN patients.

DETAILED DESCRIPTION:
Trigeminal neuralgia is a neuropathic facial pain condition which is characterised by unilateral paroxysmal pain which is excruciating, short lasting in the distribution territory of trigeminal nerve.(1) Trigeminal neuralgia is oro-facial pain restricted to one or more divisions of the trigeminal nerve. With the exception of Trigeminal Neuralgia caused by Multiple sclerosis, the pain affects one side of the face. It is abrupt in onset and typically lasts only a few seconds (2 min at maximum).Patients may report their pain as arising spontaneously, but these pain paroxysms can always be triggered by innocuous mechanical stimuli or movements. Patients usually do not experience pain between paroxysms. If they do report additional continuous pain, in the same distribution and in the same periods as the paroxysmal pain, they are considered to have Trigeminal Neuralgia with continuous pain. (IASP)(1) Trigeminal neuralgia is mainly classified into three diagnostic categories i.e. Classical, Secondary and Idiopathic. This classification is mainly based on the etiology & pain characteristics. The etiology of Trigeminal Neuralgia is not well understood, but various theories such as Compression of sensory root of trigeminal nerve by arteries & bony exostoses.(4) ,focal demyelination of trigeminal afferents near the entry of the trigeminal root into pons(2)and alteration in the central neural function followed by injury to peripheral nerves (4) are widely accepted.

Trigeminal Neuralgia has a profound effect on quality of life of the patient & expenditure on health (4). Due to the severe intensity of pain, patients avoid touching face, washing face, thus making patient's life disturbing & miserable. Even after so many years of research, it is still a challenge to treat patients suffering from Trigeminal Neuralgia. Treatment can be sub- divided into pharmacological & invasive therapies .

The pharmacological therapy include drugs such as carbamazepine ( 200-1200mg) , oxcarbazepine (300-1800mg) , lamotrigine, Gabapentin , baclofen, eslicarbazepine, sumatriptan, vixotrigine. The pre- surgical procedures like botulinium toxin A & intranasal non-inhaled CO2 have also been sporadically used (1).

A review study discussing the pharmacological options to treat trigeminal neuralgia concluded that carbamazepine & oxcarbazepine are the first choice of drugs(1). Oxcarbazepine showed equal efficacy in reducing pain attacks with better tolerability & less side effects (1) .

A recently conducted study found that carbamazepine is associated with serious side effects including CNS disturbances, somnolence, unbalance, thrombocytopenia, increase level of transaminases while OXC showed similar efficacy with less side effects. CNS disturbances encountered in patients on CBZ were triple to those on OXC & withdrawal from the treatment was also more in patients on CBZ(27%) than on OXC (18%)(12).

OXC has contemporarily been used as monotherapy in epileptic patients (8) & has proven efficacy over the CBZ. In trigeminal neuralgia, though various studies have shown that OXC produce lesser side effects, but none of the studies have compared the efficacy of carbamazepine with oxcarbazepine .

Thus the present study intends to compare the efficacy of oxcarbazepine with carbamazepine as monotherapy in patients suffering from trigeminal neuralgia.

ELIGIBILITY:
INCLUSION CRITERIA:

* Clinically proven cases of primary trigeminal neuralgia.
* Patients who are willing to participate in the study.

EXCLUSION CRITERIA:

* Intolerance to either of the two drugs
* Medically compromised patients
* Patients with pacemaker
* Patients who have previously undergone surgical treatment for TRIGEMINAL NEURALGIA.
* Patients who are already on pharmacotherapy for TRIGEMINAL NEURALGIA.
* Seizure disorder/ pregnant/ lactating
* Renal/ hepatic impairment
* History of hyponatermia
* Concurrent medication- dilantin, phenytoin

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | 10 weeks
  Visual analog scale ( scale 0 to 10, where higher score means worst outcome)

SECONDARY OUTCOMES:
Adverse effects of drugs in both the groups. | 10 weeks
  side effects will be asked at each visit
Need for adding 2nd line therapy in both the groups. | 10 weeks
  if pateint is not satisfied with treatment, then 2nd line drug will be used
Number of patients withdrawal from study due to non compliance to drug | 10 weeks
  Drug tolerability in both the groups
Treatment satisfaction in both the groups. | 10 weeks
  likert scale is used in both groups 1-5 scale, higher score means better outcome
Quality of life in both the groups. | 10 weeks
  Oral health impact profile 14 score will be used, higher score means worst outcome

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - PGIDS, Rohtak, Haryana
  - Post Graduate Institute of Dental Sciences, Rohtak, Haryana